CLINICAL TRIAL: NCT03802981
Title: Thoracic Surgery Oncology Group (TSOG) Protocol: Registry Trial of Active Surveillance for Multifocal Ground Glass Opacities (GGOs)
Brief Title: A Registry for Patients With Multifocal Ground Glass Opacities (GGOs)
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Brigham and Women's Hospital (Other); Duke University (Other); Mayo Clinic (Other); Université de Montréal (Other); University of Pittsburgh (Other); University of Toronto (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 18-541
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Ground Glass Opacities (GGOs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry study is to actively monitor people with GGOs and collect information about them, so that investigators can learn more about these lesions and about the risk of developing lung cancer in study participants whose GGOs are being monitored in the active surveillance program.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Have two or more GGOs on initial CT imaging
* GGOs must be measure ≤3.0 cm and ≥0.6 cm in the greatest dimension
* GGOs must be greater than half ground glass

A biopsy is not necessary for inclusion in the trial. Biopsy of a GGO, even with a diagnosis of adenocarcinoma, does not necessarily preclude enrollment in this surveillance protocol. In other words, patients with a diagnosis of adenocarcinoma are still eligible, at the discretion of the clinician and/or investigator, if they meet the above criteria.

Exclusion Criteria:

* Patients who are actively undergoing lung cancer treatment or have a history of lung cancer, except for cases of completely resected pathologic stage IA nonsmall cell lung cancer (NSCLC). Patients with stage IA NSCLC and multiple GGOs can enroll in this active surveillance protocol after complete resection of the NSCLC and confirmation of stage on final pathologic assessment.
* The presence of any solid lesion ≥0.6 cm suspicious for malignancy.
* Patients who are actively undergoing treatment for other malignancies

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GGOs or mixed subsolid pulmonary nodules may be recruited from participating Thoracic Oncology Surgical Group (TSOG) sites, in accordance with local institutional practice and referral patterns, and assessed for eligibility based on the criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
lung cancer-specific survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James Huang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (32):
- United States (29):
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center (Data collection only), Stanford, California
  - Hartford Healthcare, Hartford, Connecticut
  - Rush University Medical Center (Data collection only), Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - George Washington University School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute (Data Collection Only), Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Baylor University Medical Center, Houston, Texas
- Canada (3):
  - McMaster University (Data Collection Only), Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm